# Teacher Consent to Main Study

Laura Sosinsky
Principal Investigator
Telephone #: 267-350-7693
Email: Isosinsky@phmc.org

Public Health Management Corporation Centre Square East 1500 Market Street, 15th Floor Philadelphia, PA 19102



# Public Health Management Corporation Voluntary Consent to be in a Research Study

Name of Study: Sesame Street Growing Together Study

#### **Important Things to Know About This Study**

- We are asking you to be in a research study. Your participation is voluntary. If you check
  the box below, you are agreeing to be in this study. You should not check the box below
  unless you are sure you want to be in this study and all of your questions about this study
  have been answered.
- The purpose of this study is to learn more about the impact of the Sesame Street resources on teachers' and parents' knowledge, attitudes and self-reported behavior regarding family engagement, as well as the impact of the resources on children's social emotional skills (as reported by teachers and parents).
- If you agree to be in this study, you will be asked to complete surveys over a ten week
  period. You will be asked to complete baseline and follow-up teacher surveys and baseline
  and follow-up surveys for up to six of your students.
- This study involves very few risks. We have plans in place to lower these risks.
- You may not benefit from being in this study.
- We will get information about you for this study. We have plans in place to keep your information confidential.
- This form will explain all of this to you in more detail.

#### 1. What is the purpose of this study?

Public Health Management Corporation (PHMC) is doing this study to learn more about the impact of the Sesame Street's *Growing Together* online professional development course and its related-resources. Topics covered in the Growing Together course include strategies to support all areas of children's development, including children's approaches to learning (such as attention, motivation, and persistence), social skills and emotional development, language and literacy, and physical development. Specifically, PHMC is interested in the effect of the course and resources on teachers' and parents' knowledge, attitudes and self-reported behavior regarding family engagement, as well as the impact of the resources on children's social emotional development (as reported by teachers and parents).

# 2. Who is in charge of this study?

Dr. Laura Sosinsky at PHMC is in charge of this study.

## 3. Why am I being asked to be in this study?

We are asking you to be in this study because you work as a lead teacher of a classroom with at least 3 four year olds in a center whose director has agreed for the center to participate in the study.

# 4. Who will be in this study?

People from 185 childcare centers will be asked to be in this study. Up to 185 teachers will be in this study. One teacher will be from this site. Some parents will be asked to be in this study if their child's teacher is in the study.

# 5. How long will I be in this study?

You will be in this study for about three months, January - April 2020.

# 6. What are you asking me to do?

If you agree to be in this study, you will be asked to:

- 1) <u>Complete surveys</u>. You will be asked to complete 2 teacher surveys about your background, relationship with your students' parents, self-efficacy, and classroom activities. You will also be asked to complete between 6 and 12 child surveys about some of your students' social-emotional development, learning behaviors, and school readiness skills. These surveys will be done online. You will be asked to complete the baseline teacher survey and set of student surveys shortly. You will be asked to complete the follow-up teacher and students surveys in April. Each teacher survey will take about 12 minutes. Each student survey will take about 6 minutes.
- 2) Give us some personal information. We will ask for:

- A) Name
- B) Gender
- C) Race/ethnicity
- D) Age
- E) Highest Level of Education, type of degree
- F) Experience in early childhood education
- G) Name of employer
- H) Job title

We will use this information to describe the people in this study as a group.

3) <u>Be randomly assigned to the intervention (Group A) or comparison (Group B) group.</u>
Random assignment is like flipping a coin. It makes each person have an equal chance of being in each group. You and the research team do not decide which group you are in.
The intervention group (Group A) will take Sesame Street's Growing Together online course and engage in its recommended activities.

4)

# A) If you are in **Group A**, you will:

- Complete the surveys mentioned above
- Enroll in the online course and complete one unit every two weeks. The
  course includes short videos, short materials to read and printables. You
  will receive emails for every unit with specific tips and strategies to put
  into practice what you have learned in the course with children and
  families.
- Engage in the course-suggested activities with parents and students
- Completing course and engaging in course-suggested activities will take about 1.5-2.5 hours of your time each week.
- · Complete feedback forms/checklists every other week
- · Complete a program feedback form
- Participate in a telephone focus group, if invited

# B) If you are in **Group B**, you will:

- Complete the surveys mentioned above
- Engage in business-as-usual
- <u>5) Give us your contact information</u>. We will ask for your email address We will use this information to send you the online surveys. If you are assigned to Group A, we will share your name and email address with Sesame Street so that Sesame can email you newsletters and track your participation in the course.
- 6) Potentially be in a focus group. Some teachers in Group A will be invited to participate

in a focus group. A separate consent form will be given to you if you are invited.

#### 7. Will my information be kept confidential?

Yes, we will do our very best to keep your personal information confidential. We cannot promise total confidentiality. We have done several things to protect your information:

- 1. We will only share your information with people who need to use it for this study. If you are in Group A, we will share your email address with Sesame Street program staff so that Sesame can send you newsletters and resources related to this program and track participation. We will not share any information you provide to us from surveys with Sesame Street staff.
- 2. Any information kept on a computer will be in a password-protected file. Only research staff on this study will know the password.
- 3. Your research records will not have your name on them. We will use a code number instead. The code number will be kept secure and separate from your name. Only research staff on this study will have access to the code numbers and names.

<u>Exceptions to confidentiality</u>. There are times when we will break this confidentiality agreement with you:

- 1. Any information about child abuse or intent to harm self or others <u>will</u> be reported to authorities, as required by law.
- 2. We will also break this agreement if you are having a medical emergency, or if your safety is at risk.

# 8. Will my research information be used or shared for future research studies?

We will keep information that can identify you (like your name) secure and separate from your research information. We may use or share your research information (without information that can identify you) for future research studies. If we do, then we will not ask you for permission again.

# 9. What are the possible risks of being in this study?

This study involves the following risks:

1). <u>Some parts of this study may make you feel uncomfortable</u>. You may feel uncomfortable during the surveys.

To lower the risk, you can skip any survey questions you do not want to answer.

2). There may be a breach of confidentiality. We will do our best to keep your information confidential. It is still possible that your information may be seen or heard by someone who should not see or hear it.

We have taken these steps to lower this risk:

- All survey data will be collected electronically via SurveyGizmo. SurveyGizmo includes security features such as data encryption, firewalls, and secure SSL links to surveys. Electronic data will be transferred using a secure web-based server system.
- All electronic information will be kept in a password-protected computer. Only research staff on this study will know the password.

#### 10. What are the possible benefits of being in this study?

You may not get any benefits from being in this study. This study may help you with strategies for working with your students and parents, but we cannot promise this will happen. The information we get from this study may help us find ways to help children and improve the course for the future.

#### 11. Do I have to pay to be in this study?

No, you do not need to pay anything to be in this study. The course we are testing is free.

#### 12. Will I be paid for being in this study?

We will pay you for completing study tasks. In total, you can earn at most \$146 in Amazon.com gift cards and may win a tablet/Chromebook for completing these tasks:

- You will receive \$10 Amazon.com gift card for completing a baseline teacher survey
- You will receive \$8 Amazon.com gift card for completing each baseline student survey for up to six students
- You will receive \$15 Amazon.com gift card for completing a follow-up teacher survey
- You will receive \$8 Amazon.com gift card for completing each follow-up student survey up to six students
- If you complete all baseline and follow-up surveys, you will be entered into a drawing for a chance to win one of 4 tablets/Chromebooks. Your chance of winning will be at least 4 in 185
- You will receive \$25 Amazon.com gift card for completing all five feedback forms/checklists (only if you are in Group A)

For example, a comparison teacher who has the parents of five children in the study and completes all surveys at baseline (teacher survey + five child reports), but only the teacher survey and two child reports at follow-up would earn \$81 in Amazon.com gift cards and would not be entered into the drawing.

You will be paid for the baseline teacher and student surveys that you have completed by week three of the study. You will be paid for the follow-up surveys and any feedback forms that you have completed by two weeks after the study has ended. You will be paid with Amazon.com gift cards via email. If you drop out of the study or are asked to leave the study, you will still be able

to keep the money you are given.

#### 13. Do I have to be in this study?

No, you do not have to be in this study. No one will treat you differently if you do not want to do this. You will not get in trouble if you do not want to be in this study. If you do not want to be in this study, tell us and do not check the box below. If you want to be in this study, tell us and check the box below.

You can say "yes" now and change your mind later. If you do not want to be in this study anymore, you can tell Dr. Laura Sosinsky. Dr. Sosinsky is the Principal Investigator (the person in charge of this study). Dr. Sosinksy's phone number is 267-350-7693 and her email address is Isosinsky@phmc.org. You can ask us to get rid of all of your study information.

# 14. What other choices do I have if I choose not to be in this study?

If you do not want to be in this study, you can still access the Growing Together course by going to:

https://sesamestreetincommunities.org/professional-development/courses?training=growing-together

# 15. Can I be asked to leave this study?

We may ask you to stop being in this study if you stop working in your current classroom at your current center. We will notify you via email if we remove you from the study. The data gathered up until that point will be kept and will remain confidential.

You cannot be in this study if you are no longer working as a lead teacher of a classroom with at least 3 four year olds in a center whose director has agreed for the center to participate in the study.

# 16. Will I be contacted in the future about this study?

We will contact you in the future if:

- There is new or important information that may make you change your mind about being this study.
- We learn important information about your health, safety, or rights after the study ends.

We will not contact you for any other reason.

#### 17. Who can I call about my rights as a participant in this research study?

The Institutional Review Board (IRB) makes sure that this study is being done right. You can call the PHMC IRB at 1-800-335-9875 or email ResearchCompliance@phmc.org if:

- You have questions about your rights as a study participant.
- · You want to make a complaint about this study.
- You get an injury from being in this study.

If you have questions about this study, you can contact Dr. Sosinsky. Dr. Sosinsky's phone number is 267-350-7693 and her email address is Isosinsky@phmc.org.

18.

#### **Documentation of Consent**

- I have read, or been read, this form.
- All of my questions were answered.
- I understand why this study is being done and what I will be asked to do.

0%

- I agree to be in this study.
- I will get a copy of this form to keep.

| Please indicate that you have read the above information. * |
|---|
| I have read the above information. |
| 19. Your Full Name: * |
| 20. Your Email: (Please share an email that you will be checking regularly and using for the study.) |
| Submit |